CLINICAL TRIAL: NCT06312644
Title: Observational Study of Ultomiris® (Ravulizumab) Safety in Pregnancy
Brief Title: Study of Ultomiris® (Ravulizumab) Safety in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D9289C00007
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ultomiris-exposed Pregnant/ Postpartum; Pregnancy; Paroxysmal Nocturnal Hemoglobinuria (PNH); Atypical Hemolytic Uremic Syndrome (aHUS); Generalized Myasthenia Gravis (gMG); Neuromyelitis Optica Spectrum Disorder (NMOSD)
Keywords: Ultomiris; pregnancy; PNH; aHUS; gMG; NMOSD
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Atypical Hemolytic Uremic Syndrome; Myasthenia Gravis; Neuromyelitis Optica | interventions — ravulizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ultomiris — Participants exposed to Ultomiris at any point during the 40 weeks prior to conception (LMP+14 days) or at any point during pregnancy or breastfeeding up to 52 weeks after birth.
  Other Names: There is no interventional drug. Ultomiris treatment is an inclusion criterion.

SUMMARY:
The primary objective of this study is to describe the frequency and characteristics of pregnancy outcomes and maternal complications among participants exposed to Ultomiris and to describe the frequency and characteristics of selected fetal/neonatal/infant outcomes in utero, at birth, and through 1 year of age after exposure in utero or via breastmilk.

DETAILED DESCRIPTION:
This observational study will collect prospective and retrospective data in participants exposed to Ultomiris during pregnancy and/or breastfeeding to assess risk of maternal complications, adverse effects on the developing fetus, and adverse effects on the infant.

ELIGIBILITY:
Inclusion Criteria:

* Female participant must have a medically confirmed qualifying pregnancy (prospectively or retrospectively identified).
* Participant informed consent (written or e-consent per local regulations or ethics committee requirements) must be obtained prior to the participant's enrollment. If the participant is a minor, consent must be obtained from the parent or legal guardian, with assent from the minor (as locally appropriate).
* Willing to provide contact information for the participant.
* Willing to authorize HCP(s) to release maternal and infant medical information to the study, upon request, if applicable to current local regulations.
* Diagnosed with an indication for which Ultomiris is approved, based on HCP or medical records.
* Exposed to Ultomiris at any point during the defined exposure window based on HCP or medical record documentation. (If exact exposure dates are unknown, the reporter must be able to specify or estimate trimester or timing of exposure [prior to conception as LMP+14 days, or during breastfeeding].)
* Use of Ultomiris per local product information (i.e., United States Prescribing Information [USPI] or summary of product characteristics [SmPC])

Exclusion Criteria:

* Participants who are unable to provide consent or assent (as locally appropriate) (e.g., diagnosed with severe psychiatric conditions or severe intellectual disabilities) will be excluded from this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants exposed to Ultomiris at any point up to 40 weeks prior to conception (Last Menstrual Period +14 days) through pregnancy and/or breastfeeding through the first 52 weeks of the infant's life.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2034-07-11 (Estimated); Study Completion 2034-07-11 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Complications | Up to 4 weeks post-delivery
  Pregnancy outcomes
Maternal Complications | Up to 4 weeks post-delivery
  Maternal Complications may include pre-eclampsia, eclampsia, deep-vein thrombosis (DVT), pregnancy-induced hypertension, gestational diabetes, preterm labor, placenta previa, and postpartum hemorrhage
Fetal/Infant Outcomes | In utero through 52 weeks of age after exposure to Ultomiris (in utero or via breastmilk)
  Fetal (in Utero)/infant (for Live Born Births) may include major congenital malformation (MCMs), full-term birth, preterm birth, low birth weight, size for gestational age, neonatal death, perinatal death, infant death, serious and severe infections of infants, infant hospitalization, growth delays, and abnormal postnatal growth and development

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Williams, Principal Investigator — North American Coordinating Center (NACC)
Locations (7):
- Research Site, Boston, Massachusetts, United States
- Research Site, Melbourne, Victoria, Australia
- Research Site, Paris, France
- Research Site, Essen, Norte-Westfalia, Germany
- Research Site, Rome, Italy
- Research Site, Seoul, South Korea
- Research Site, London, United Kingdom